CLINICAL TRIAL: NCT04297514
Title: Effects of Pulmonary Rehabilitation According to Gender, in COPD Patients
Brief Title: Effects of Respiratory Rehabilitation by Gender in COPD Patients
Acronym: REHABGENRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: REHABGENRE (29BRC20.0030)
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2022-08

CONDITIONS: COPD; Pulmonary Rehabilitation
Keywords: COPD; pulmonary rehabilitation; Dyspnea; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Without calling into question the effectiveness of pulmonary rehabilitation in women, the difference in outcome by gender was not established due to insufficient evidence .

Studies demonstrating the effectiveness of pulmonary rehabilitation include a majority of men, which no longer corresponds to the sex ratio of the disease. The impact of gender on pulmonary rehabilitation outcomes was not established due to insufficient evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* No opposition filed
* Patient with COPD
* Completed participation in respiratory rehabilitation program

Exclusion Criteria:

* Refusal of participation
* Patient under tutorship or curatorship
* No final assessment
* Patients with sex changes in marital status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients undergoing a pulmonary rehabilitation program
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
DYSPNEA-12 | Change from baseline Dyspnea-12 score at 4 weeks
  Dyspnea-12 allows to evaluate sensori and emotional dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PhD, Principal Investigator — CH des pays de Morlaix
Locations (1):
- CH des pays de Morlaix, Morlaix, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 Months and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.